CLINICAL TRIAL: NCT03090867
Title: Participation of Relative or Surrogate in the Patient's Care in Reanimation
Acronym: PARTICIPATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ICAN Nutrition Education and Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P150301
Record Dates: First submitted 2017-02-06; First posted 2017-03-27 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Critical Care; Anxiety Depression
Keywords: Clinical Practice Guideline; Critical care; Family-centered care; Professional-family relations; Family nursing; Anxiety; Depression; Participation in care
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional arm (Active Comparator): The relative or surrogate will not be encouraged to perform care. The management of the relative or surrogate wi ll not changed from the regular standard of the ICU.
  Interventions: Other: Conventional ,care
- The relative/surrogate will be encouraged to perform care (Experimental): The relative or surrogate will perform at least two cares a week . A manual will be given to the relative or surrogate, explaining the different care he can choose to perform on the patient.
  The care proposed are: feeding, mouth care, hair wash, shaving, eye care, hand, foot and face massage.
  All care are planned and perform under the supervision or/and in collaboration with a caregiver.
  Each care is written down on a collecting sheet.
  Interventions: Other: Relatives or surrogates are encouraged to perform care

INTERVENTIONS:
Other: Relatives or surrogates are encouraged to perform care — The relative or surrogate will perform at least two cares a week among feeding, mouth care, hair wash, shaving, eye care, hand, foot and face massage.
  All care are planned and perform under the supervision or/and in collaboration with a caregiver.
  The relative or surrogate will give his opinion by completing the study questionnaires.
  Arms: The relative/surrogate will be encouraged to perform care
Other: Conventional ,care — The relative or surrogate will not be encouraged to perform care. The management of the relative or surrogate wi ll not changed from the regular standard of the ICU.
  Arms: Conventional arm

SUMMARY:
ICUs have always perceived by the public has a very technical unit with a restricted and/or forbidden access. Physical alteration of the patient, seeing the patient sedated, the large numbers of devices, the alarms and an uncertain prognosis. All this factors can be perceived by people close to the patient as a source of stress. In the literature, numerous studies have shown that families develop anxiety and depression symptoms while their loved one is hospitalized in the ICU. French intensive care societies thought of ways to prevent or diminish these symptoms. The 6th consensus conference on " Live better in the ICU " recommends: effective and adapted information, large visiting hours to reach an unrestricted access and family participation in care.

The unit has taken this path to improve patient and family centered care by: creating a welcome leaflet, a room dedicated to meetings with families and an ICU open 24/7bto families, with the possibility for children to visit their parents. Hence, spontaneously, relatives have expressed the wish to participate to certain care and when participating, expressed their satisfaction. This observation and testimonies from family members and patients led us to think about the impact of participation of care. Two major French studies have shown contradictory outcomes: 16% of families would have been willing to participate in the first study against 97% in the second one. These studies were survey done after the ICU discharge.

No study today has assessed the actual impact of family participation in care. The aim of this clinical trial is to diminish anxiety and depression symptoms. By participating in care, relatives can develop or strengthen a relationship of trust with caregivers. It could contribute also to a better understanding of the plan of care and an easier context to announce negative outcomes.

DETAILED DESCRIPTION:
Randomisation visit - D1:

After checking the eligibilities criteria, a member of the staff will explain to the patient and his relative or surrogate the purpose and the planning of the study. The inform consent will be signed by the physician of the study. Two informs consents will be signed : one by the patient and the other one by the relative or surrogate. The randomisation will be done after collecting these consents.

After the draw, the subjects will be randomized either in the control group "Conventional support" or the experimental group "Intervention".

Questionnaires to be completed by the :

* relatives or surrogates: Hospital Anxiety and Depression scale (HAD scale), Multidimensional Fatigue Inventory (MFI20), Zarit Burden Interview (ZARIT sale) , Beck Depression Inventory (Beck), State-Trait Anxiety Scale (STAI) and "preliminary"
* patient if possible: HAD scale

Admission + 10 days visit:

Questionnaires to be completed by the relatives or surrogates: HAD scale, MIF20, ZARIT, Beck, STAI and "discharge"

ICU discharge visit :

Questionnaires to be completed by the :

* relatives or surrogates: HAD scale, MIF20, ZARIT, Beck, STAI and "discharge"
* patient if possible: HAD scale

Medical staff:

In order to evaluate the feeling of the ICU staff, a satisfaction questionnaire will be propose at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion criteria

1. An adult related to the ICU patients, giving his written consent to participate to the study
2. Being present at the patient's bedside at least twice a week
3. Speaking and writing comprehension of the french language
4. Adult ICU patient, admitted in the ICU for less than 72 hours, whatever its pathology
5. Predictable ICU stay over a week

Exclusion criteria

1. Refusal of the relative or surrogate
2. Refusal of the patient
3. The relative or surrogate can't be present at the patient's bedside at least twice a week
4. Relative or surrogate already participating in the care of the patient for a chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HAD scale at ICU's discharge | From baseline and at the patient's discharge from the ICU assessed up to 3 months
  HAD Scale : The primary outcome measure is the relative or surrogate HAD (Hospital Anxiety and Depression Scale) score evolution.
  The expected result is a reduction by two points of the total HAD score through active participation in care.

SECONDARY OUTCOMES:
Evolution of the relative or surrogate anxiety/depression | at baseline and after 10 days of ICU hospitalization.
  The relative or surrogate will complete the HAD scale and other anxiety/depression questionnaires.
Evolution of the relative or surrogate anxiety/depression | at baseline and at ICU's discharge assessed up to 3 months
  The relative or surrogate will complete the HAD scale questionnaires and anxiety/depression questionnaires.
Evaluation of the satisfaction's relatives or surrogates regarding their participation in the ICU patient care by a questionnaire | At the patient's ICU discharge assessed up to 3 months
  Concern different aspects of the patient's management: listening skills and support from the ICU team, medical information about the patient, benefits and difficulties encountered while participating in care
Evaluation of the satisfaction of the ICU staff by a questionnaire | Through study completion an average of 12 months
  Evaluate the feeling of the ICU staff regarding participation in care of surrogates and assess its evolution at the end of the study.
  The ICU staff can describe which benefits and difficuties they encountered while caring for the patient with the relative or surrogate.
  At initiation visit and at closing of the center
Quantify which care have been realized by the relatives or surrogates | Through study completion an average of 12 months
  Each time a relative or surrogate is caring for the patient, the ICU staff will write it on a specific sheet.
  At the end of the study, all this data will be gathered to see which care have been done more often
HAD scale of the patient | At the ICU discharge assessed up to 3 months
  The patient completes the HAD scale if his mental state allows it

CONTACTS AND LOCATIONS:
Overall Officials: Alain COMBES, M.D, Ph.D, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azoulay E, Pochard F, Chevret S, Arich C, Brivet F, Brun F, Charles PE, Desmettre T, Dubois D, Galliot R, Garrouste-Orgeas M, Goldgran-Toledano D, Herbecq P, Joly LM, Jourdain M, Kaidomar M, Lepape A, Letellier N, Marie O, Page B, Parrot A, Rodie-Talbere PA, Sermet A, Tenaillon A, Thuong M, Tulasne P, Le Gall JR, Schlemmer B; French Famirea Group. Family participation in care to the critically ill: opinions of families and staff. Intensive Care Med. 2003 Sep;29(9):1498-504. doi: 10.1007/s00134-003-1904-y. Epub 2003 Jul 10. PMID 12856124
- [Background] Garrouste-Orgeas M, Willems V, Timsit JF, Diaw F, Brochon S, Vesin A, Philippart F, Tabah A, Coquet I, Bruel C, Moulard ML, Carlet J, Misset B. Opinions of families, staff, and patients about family participation in care in intensive care units. J Crit Care. 2010 Dec;25(4):634-40. doi: 10.1016/j.jcrc.2010.03.001. PMID 20435430